CLINICAL TRIAL: NCT06811675
Title: The Efficacy of Dexamethasone in Combination With N-acetylcysteine in Preventing Neurocognitive Sequelae Due to Carbon Monoxide Poisoning
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH113-REC1-201
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Carbon Monoxide Poisoning; Delayed Neurocognitive Sequelae
Keywords: Carbon Monoxide Poisoning; Dexamethasone; N-acetylcysteine; Delayed Neurocognitive Sequelae
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Dexamethasone; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone and n-acetylcysteine (Experimental): Dexamethasone 10mg IV STAT +QD for 3 days+NAC IV 200mg/kg over 4 h, then 100 mg/kg over 16 h
  Interventions: Drug: Dexamethasone and N-acetylcysteine (NAC)
- placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone and N-acetylcysteine (NAC) — Dexamethasone 10mg IV STAT +QD for 3 days+NAC IV 200mg/kg over 4 hours, then 100 mg/kg over 16 hours
  Arms: dexamethasone and n-acetylcysteine
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
Background and Aim: Carbon monoxide (CO) poisoning is a significant public health issue that can cause delayed neuropsychological sequelae (DNS). DNS mechanisms involve oxidative stress, inflammation, and immune injury. Although hyperbaric oxygen therapy is widely used, its efficacy in preventing DNS remains inconclusive. Preclinical and retrospective studies suggest that Dexamethasone (anti-inflammatory and immunosuppressive) and N-acetylcysteine (antioxidant) may reduce DNS risk. This study hypothesizes that their combination can effectively prevent DNS.

Methods: This prospective pre-post intervention study will enroll CO poisoning patients into treatment (Dexamethasone + N-acetylcysteine) and control groups. The primary outcome is the incidence of DNS within six weeks post-treatment.

Objective: To determine whether combining Dexamethasone and N-acetylcysteine reduces the incidence of DNS following CO poisoning.

ELIGIBILITY:
Inclusion Criteria:

* History and clinical symptoms consistent with CO poisoning (initial blood carboxyhemoglobin (COHb) levels >5%, or >10% for smokers).

Exclusion Criteria:

* Concurrent use of other potentially lethal toxins. Severe trauma or burns that could be fatal. No spontaneous heartbeat or blood pressure before arrival. Poisoning time exceeding 24 hours before hospital arrival. Minors (under 18 years of age). Pregnant women. Patients or their families refuse to sign the consent form. Contraindications for the use of Dexamethasone or N-acetylcysteine (such as severe allergies) or when the physician assesses the risks outweigh the benefits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delayed neurological sequelae following carbon monoxide exposure, as assessed by clinical evaluation | 2 weeks, 6 weeks, 3 months
  Questionnaire:
  Parkinson-like syndromes Concentration deficits Gait and motor disturbances Memory loss Bradykinesia Cognitive impairment Intention tremor Dementia Myoclonus Personality changes Dyspraxia Anxiety Dysphasia Extreme emotional lability Ataxia Psychosis Postural instability Depression Vertigo Mania Cortical blindness Insomnia Hearing loss, tinnitus Chorea EEG abnormalities Epilepsy Peripheral neuropathies Recurrent headaches Fecal or urinary incontinence
  Criteria:
  The presence of any delayed-onset symptoms listed above, emerging at least 2 days after initial recovery from carbon monoxide poisoning, will require confirmation by a toxicologist, neurologist, or psychiatrist experienced in diagnosing delayed neuropsychiatric sequelae (DNS) following CO exposure.

SECONDARY OUTCOMES:
Number of participants with cognitive impairment following carbon monoxide exposure, as assessed by the Mini-Mental State Examination (MMSE) | 2 weeks, 6 weeks, 3 months
  Cognitive impairment will be assessed using the Mini-Mental State Examination (MMSE) at 2 weeks, 6 weeks, and 3 months post-exposure. A score of ≥24 (out of 30) indicates normal cognition, while lower scores indicate varying degrees of impairment: mild (19-23), moderate (10-18), and severe (≤9). The number of participants meeting the criteria for cognitive impairment will be recorded at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No